CLINICAL TRIAL: NCT00276991
Title: Modest Phase 1 and Phase II Clinical Studies on Traditional CAM Therapy in the Treatment of HIV/AIDS
Brief Title: Traditional CAM Therapy in the Treatment of HIV/AIDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding prevented the recruitment of 1000 HIV Patients all over India
Sponsor: Traditional Alternative Medicine Research, India (Other)
Responsible Party: Principal Investigator, RAMAKRISHNAN MADHUSOODANAN, Director, Traditional Alternative Medicine Research Center TAMRC-INDIA., Traditional Alternative Medicine Research, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAM10; NCT00385424 (obsolete NCT alias); NCT00505193 (obsolete NCT alias); NCT00554060 (obsolete NCT alias)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: HIV Infections
Keywords: Prolonged Viral Suppression; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- "Kallunk oxide (Immunotherapy)" (Other): The participants were received a daily regimen of "Kallunk oxide(Immunotherapy)" .
  Interventions: Drug: "Kallunk oxide (Immunotherapy) "

INTERVENTIONS:
Drug: "Kallunk oxide (Immunotherapy) " — The study was assigned only one Arm >450 cu/mm^3 of baseline CD + T cells. HIV type-1 subjects were received one drug, a daily regimen of "Kallunk oxide(Immunotherapy) + Long Pepper", that is a combination of a traditional alternative medicine(Complementary and Alternative Medicine CAM) as "Kallunk oxide" and appropriate drug carrier antidote. The drug assigns to 0.100 mg and 0.200 mg "Kallunk oxide" molecules with 199.900 mg, and 499.800 mg "Antidote"( This antidote was used as a carrier of "Kallunk oxide" molecules), respectively, for children and adults. Dosage: 200 mg for children and 500 mg for adults. This powder form sample size product was administered once daily dose on 5 days treatment. The Botanical name of the antidote is "Piper Longum".
  Other Names: 'Kallide'

SUMMARY:
This research work is important for the cure/control of HIV infection. The objectives of a treatment case on HIV patient is essentially to bring down the viral load closer to undetectable level. The studies are depend on the potential influence of 'Kallunk Oxide' on the CD4+ T cells and the effectiveness on surface of HIV-1. The basic study is to break surface protein and directly inhibit a protein's increased functions, not only in the CD4+T cell but also CD3 and CD8+ T cells, by appropriate antidote.

The 'Yogaprabhava', the drug's effectiveness, and progressive immunity with diet and lifestyle can be more easily studied.

DETAILED DESCRIPTION:
This research was individual investigator initiated meritorious project to identify potential roles for the safe and effective use of Complementary and Alternative Medicine CAM in the treatment of HIV infection.

This modest Phase-I and phase II clinical trials were intervention Studies. In the case of HIV infections, these studies were formulated each 20 random numbered batch. The Principal Investigator (PI) selects the informed consented patients and the recruited study was adhered by Helsinki Declaration.

Selection of subjects: HIV patients with CD3, CD4, and CD8 + T cell counts >450 cu/mm^3 were enrolled in Wing No: 1 group. HIV patients with CD+ T cell counts >450 cu/mm^3 were recruited for basic Arm study. The selected Arm - 1 of this research, the specific and potential milestone on baseline CD+T cell counts >450 cu/mm^3 was determined from the outcomes of previously conducted Observational Phase-1 study data.

The statistical evaluation laboratory on parameters in exists group was measured through Immune Cells Count Assay. The prolonged viral suppression and reversal of HIV seropositivity were the ultimate research outcomes and this study was evaluated the safety and efficacy of this drug. Absolute assays of Viral Load, Lymphocyte Enumeration, Western Blot blood test and convinced mean values and reference range methods were adopted for laboratory study.

The drug was administered as optimal doses 200 mg and 500 mg to study subjects, respectively, between 8 and 17 years old children and 18 and 65 years old Men and Women as anticipated 500 Female and 500 Male participants. The ELISA/P-24 test was used to confirm HIV-seropositivity.

The patients safe and effective optimum dose was the primary out come measure and the Viral Load assay and Immune Cells Count assay were the secondary outcome measure.

The randomized numbers were arranged with single patient's clinical records. Patient's body weight, CD4 T cells count, skin thickness, body measurements, blood pressure, temperature, pulse rates, anti body count, and other hematological examinations were investigated before and after the treatment period.

The well-designed research team minds the symptoms such as nausea, fatigue,weight loss, sweating, shortness of breath, joint pain etc and the Side effects of this treatment, if any, could be carefully noted. On entry and at the end of this study, the biochemical investigations such as urine examination, serum lipoprotein and cholesterol were individually noted.

Patient's temperature, digestion complaints, or chill, etc could treated by medicine and restricted diets without using mutton soup, milk, and cow ghee. The study was reduced patient's stress as well as depression and also managed the productivity, emotional well being, immunity and quality of life by the practice of this treatment.

The study was handled a transparent privacy environment to recruit HIV-infected people in India.

Dosage:

HIV patients were administered with once daily dose of sample size product, 500 mg for adults and 200 mg for children (up to 8 years old), as one course.

Controlled Nourished diet:

All patients were adhered with nourished diet protocol. The controlled diets were milk (only 1/2 cup), rice and wheat food products, cow ghee, green gram, mutton soup, and prepared black pepper added vegetable foods.

Restriction:

HIV-Patients were not used salts, other oils, mustard, and tamarind fish items within 10 days of this medication use.

Drug Administration:

HIV- patients were used one drug "Kallunk oxide (Immunotherapy)" as calcined/or oxidized molecules. The powder form sample size medicine was put into 1/2 cup hotter water (an adjuvant).

Precaution:

No precautions be needed. Patients were not used sediments at the bottom of the cup.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV/AIDS
* Able to swallow tablets or powder form medicine
* Able to eat nutritional foods
* HIV infected patients
* Signed consent of parent or guardian for patients under 21 years of age
* Interest to use of study drugs
* Follow at a participating clinical site and
* Children of any age (greater than 8 years old)

Exclusion Criteria:

* Medical side effects
* Pregnant or breast feedings
* History of significant cardiac abnormalities or dysfunction
* Anti Retro viral Treatment ART used patients
* Received certain drugs or treatments
* Unable to followed at a participating clinical center
* Children less than 8 years old
* Any serious conditions (severe chronic stage AIDS cases) at study entry that may affect the results of the study.
* Allergy to any of the study drugs or their formulations
* Tobacco using patients
* Alcohol using patients and
* Drug addicting patients.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
SafeDose, | Six months follow up

SECONDARY OUTCOMES:
Viral Load Assay | Three months follow up
Absolute Immune Cells Count Assay(CD3, CD4, and CD8 + T cells) | Three months follow up in Phase - II study
Prolonged Viral Suppression | Six Month's Follow up study( In Phase-II Study)

CONTACTS AND LOCATIONS:
Overall Officials: Ramakrishnan Madhusoodanan, PHD, Principal Investigator — Traditional Alternative Medicine Research Center
Locations (1):
- Project Site Office, Hospital of Integrated Research Site HIRS(New), Ahammed Nagar, Mathura Nagar, Bhingar- PO, Mumbai, India